CLINICAL TRIAL: NCT07238283
Title: Irinotecan Hydrochloride Liposome Injection (II) in Combination With Oxaliplatin, 5-fluorouracil, Calcium Folinate Versus Nab-paclitaxel in Combination With Gemcitabine for First-line Treatment of Metastatic Pancreatic Cancer: an Open, Randomized, Multicenter Phase III Trial.
Brief Title: Irinotecan Hydrochloride Liposome Injection (II)in Combination With Oxaliplatin, 5-FU/LV Versus AG for First-line Treatment of Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR070803-308
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: First-line Treatment of Metastatic Pancreatic Cancer
MeSH Terms: interventions — Oxaliplatin; Fluorouracil; Leucovorin; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): Irinotecan Hydrochloride Liposome Injection (II) in combination with oxaliplatin, 5-fluorouracil, calcium folinate
  Interventions: Drug: Irinotecan Hydrochloride Liposome Injection (II); Oxaliplatin; 5Fluorouracil; Calcium folinate
- Treatment group B (Active Comparator): nab-paclitaxel in combination with gemcitabine
  Interventions: Drug: nab-paclitaxel; gemcitabine

INTERVENTIONS:
Drug: Irinotecan Hydrochloride Liposome Injection (II); Oxaliplatin; 5Fluorouracil; Calcium folinate — Irinotecan Hydrochloride Liposome Injection (II) in combination with oxaliplatin, 5-fluorouracil, calcium folinate
  Arms: Treatment group A
Drug: nab-paclitaxel; gemcitabine — nab-paclitaxel in combination with gemcitabine
  Arms: Treatment group B

SUMMARY:
This study is a randomized, open-label, multicenter Phase III clinical trial designed to evaluate the efficacy and safety of Irinotecan Hydrochloride Liposome Injection (II) combined with oxaliplatin and 5-FU/LV versus nab-paclitaxel combined with gemcitabine as first-line treatment for advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status 0 or 1
2. Histological or cytologically confirmed pancreatic cancer that has not been previously treated in the metastatic disease.
3. Life expectancy of greater than or equal to3 months.
4. At least one measurable lesion is present according to the efficacy evaluation criteria for pancreatic cancer (RECIST 1.1)
5. Able and willing to provide a written informed consent

Exclusion Criteria:

1. Patients with pancreatic cancer originating from extrapancreatic ductal epithelium, including pancreatic neuroendocrine carcinoma, acinar cell carcinoma of the pancreas, pancreatoblastoma, and solid-pseudopapillary tumor;
2. Known history of central nervous system (CNS) metastases.
3. Severe infection (> CTCAE grade 2), such as severe pneumonia, bacteremia, infection complications, etc. requiring inpatient treatment, occurred within four weeks before enrollment, and symptoms and signs of infection requiring intravenous antibiotic therapy (except for prophylactic antibiotics) occurred within two weeks before enrollment;
4. Patients with cardiac clinical symptoms or diseases that are not well controlled, such as: (1) Patients with NYHA class 2 and above cardiac failure; (2) unstable angina; (3) myocardial infarction that occurred within 6 months; (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 662 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From study start until target OS events have occurred (approximately 18 months after last patient enrollment)

SECONDARY OUTCOMES:
Objective Response rate (ORR) | up to 6 months following the date the last patient was randomized
  ORR is defined as the percentage of participants who have a best overall response of complete response (CR) or partial response (PR), per RECIST 1.1.
Disease Control Rate | up to 6 months following the date the last patient was randomized
  The study is designed to evaluate the disease control rate with advanced pancreatic cancer. DCR is defined as the percentage of patients with a best response of CR, PR, or stable disease (SD).
Duration of Response | up to 6 months following the date the last patient was randomized
  DoR is defined as the time from first documentation of response (CR or PR whichever occurred first, as per RECIST version 1.1) to disease progression or death, whichever is earlier.
Progression free survival (PFS) | From the date of first dose of study drug until progressive disease (PD), death, whichever occurs first,assessed up to 18 months
  PFS is defined as the time from the date of first dose of study drug to the date of the first documentation of disease progression or date of death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided